CLINICAL TRIAL: NCT03909932
Title: How to Dress up in Neuro-urology Department
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Other Study IDs: GRC 001 GREEN
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Clothing
Keywords: Physician attire; neuro-urology; urodynamic; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients enrolled in the cross-sectional study: Patients over 18 years old, consulting in neuro-urology department.
  Interventions: Other: Observational study : no intervention

INTERVENTIONS:
Other: Observational study : no intervention — Observational study : only exporting data

SUMMARY:
This study assess patient preferences and perceptions regarding physician dress code in a neuro-urology department.

DETAILED DESCRIPTION:
Patient satisfaction with care contribute to therapeutic compliance and adherence leading to better outcomes.Various factors impact on patient satisfaction as communication with nurses and doctors, pain management, timeless of assistance, explanation of medications administered, cleanliness of room and bathroom, discharge planning, noise level at night…ith increasingly consultation requests and delays and rushed patient-physician encounter, the ability to gain a patient's confidence to optimize health outcomes has become a real challenge. Petrilli and al. described the role of physician attire on patients perceptions and highlight its importance in patient confidence, trust and satisfaction.Therefore, targeting physician attire to improve the patient experience has become a topic of interest.

In a neuro-urology department with outpatients services and additional explorations (urodynamic, anorectal manometry, electromyographic testing), the physician attire is an outstanding issue because of this non-surgical activity but its procedural therapies.

The aim of this cross-sectional study was to examine patient perceptions and preferences regarding physician dress code in a neuro-urology department.

In this study, the investigators develop a questionnaire based on expert meetings and literature review of the role of physician attire on patient preference and satisfaction. This lead to a short questionnaire with 2 sections and 4 questions. In the first section, 3 photographs of different physician attires will be presented: casual attire with white coat, scrubs and scrubs with white coat. The face of the physician will be hidden, pose lighting and environment will be similar. Respondents will be asked to select their ideal attire and to mention if any attire shock them. The second section sought respondents' general opinions regarding physician attire, its importance and relation with patient satisfaction.

Surveys will be filled in a neuro-urology department of a university hospital in France. The questionnaire will be administered to adult patients who will be consulting or adminting for a one-day- hospitalization. The patient will fill the survey alone or with help from any relative accompanying him. The research staff will deliver and collect the completed form. Demographic data (age, sex, occupational category, education level), presence of neurological disease, patient already know of the department or first visit, reason of the external consultation or of the one-day-hospitalization will be collected.

Statistical analysis will be carried out using R 3.2.3 software (R Development Core Team, http://www.R-project.org) and R studio version 1.0.136.

Descriptive statistics (means, percentage) and SD will be used to describe the population and the responses to the questionnaire. Differences between the rating and the patients' characteristics will be assessed using analysis of variance or Chi2 tests. A p value of less than 0.05 will be considered statistically significant.

This study was approved by a local ethics committee. No identifying information was collected from those that completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Appointment in neuro-urology department

Exclusion Criteria:

* refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who were consulting in neuro-urology department
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
preference of physician dress code | 1 day
  the dress code chosen by patient

SECONDARY OUTCOMES:
perception of physician attire | 1 day
  importance of physician attire for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PHD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital tenon, Paris, France